CLINICAL TRIAL: NCT01367301
Title: A Pilot Trial of Radiation Therapy "Sandwiched" Between Paclitaxel and Carboplatin in Patients With Uterine Carcinosarcoma
Brief Title: Radiation Therapy, Paclitaxel, and Carboplatin in Treating Patients With Uterine Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual. PI left the institution
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-02-064; NCI-2013-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-089; 11-02-064 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Stage IA Uterine Sarcoma; Stage IB Uterine Sarcoma; Stage IC Uterine Sarcoma; Stage IIA Uterine Sarcoma; Stage IIB Uterine Sarcoma; Stage IIIA Uterine Sarcoma; Stage IIIB Uterine Sarcoma; Stage IIIC Uterine Sarcoma; Stage IVA Uterine Sarcoma; Stage IVB Uterine Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — Paclitaxel; Taxes; Carboplatin; Brachytherapy; Linear Energy Transfer; Therapeutics; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, radiotherapy) (Experimental): CHEMOTHERAPY (weeks 1-9, 14-22): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 14-22.
  RADIATION THERAPY (weeks 8-16): Patients undergo external beam pelvic radiation therapy once a day, 5 days a week for 5 weeks during weeks 8-13. Patients then undergo HDR brachytherapy or IMRT once weekly during weeks 14-16.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Radiation: external beam radiation therapy; Radiation: brachytherapy; Radiation: intensity-modulated radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Taxol (TAX)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Radiation: external beam radiation therapy — Undergo external beam radiation therapy
  Other Names: EBRT
Radiation: brachytherapy — Undergo HDR brachytherapy
  Other Names: low-Linear energy transfer (LET) implant therapy; radiation brachytherapy; therapy, low-LET implant
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies radiation therapy, paclitaxel, and carboplatin in treating patients with uterine cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Giving radiation with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the one year recurrence-free survival in patients with uterine carcinosarcoma treated with "sandwich" therapy-including defining the patterns of recurrence in patients with carcinosarcoma who were treated with this regimen.

II. To evaluate the toxicity and tolerability of pelvic radiation "sandwiched" between cycles of paclitaxel/carboplatin chemotherapy in patients with uterine carcinosarcoma.

III. To correlate surrogate endpoint biomarkers with progression-free survival and prognosis.

OUTLINE:

CHEMOTHERAPY (weeks 1-9, 14-22): Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 14-22.

RADIATION THERAPY (weeks 8-16): Patients undergo external beam pelvic radiation therapy once a day, 5 days a week for 5 weeks during weeks 8-13. Patients then undergo high dose radiation (HDR) brachytherapy or intensity-modulated radiation therapy (IMRT) once weekly during weeks 14-16.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented uterine carcinosarcoma with no visible residual disease
* Surgical staging to include total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, and lymph node samplings
* Patients must be entered no more than 12 weeks post operatively
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2
* Written voluntary informed consent

Exclusion Criteria:

* Serum glutamic oxaloacetic transaminase (SGOT) and /or serum glutamate pyruvate transaminase (SGPT) > 2.5 times the institutional upper limit of normal
* Total serum bilirubin > 1.5 mg/dl
* History of chronic or active hepatitis
* Serum creatinine > 2.0 mg/dl
* Platelets < 100,000/mm3
* Absolute neutrophil count (ANC) < 1500/mm3
* Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
* Patient has severe or uncontrolled concurrent medical disease (e.g. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patient with any prior chemotherapy or radiotherapy for pelvic malignancy
* Patients with any history of cancer with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the past five years
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07-08 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merieme Klobocista, Principal Investigator — Albert Einstein College of Medicine; Dennis Yi-Shin Kuo, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants were enrolled into the study between 7/08/2011-3/8/2016. Three participants screen failed prior to consenting.
Groups:
- Treatment (Paclitaxel, Carboplatin, Radiotherapy): CHEMOTHERAPY (weeks 1-9, 14-22): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 14-22.
  RADIATION THERAPY (weeks 8-16): Patients undergo external beam pelvic radiation therapy once a day, 5 days a week for 5 weeks during weeks 8-13. Patients then undergo High Dose Rate (HDR) brachytherapy or Intensity-modulated Radiation Therapy (IMRT) once weekly during weeks 14-16.
  paclitaxel: Given IV
  carboplatin: Given IV
  external beam radiation therapy: Undergo external beam radiation therapy
  brachytherapy: Undergo HDR brachytherapy
  intensity-modulated radiation therapy: Undergo IMRT
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Paclitaxel, Carboplatin, Radiotherapy): CHEMOTHERAPY (weeks 1-9, 14-22): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 14-22.
  RADIATION THERAPY (weeks 8-16): Patients undergo external beam pelvic radiation therapy once a day, 5 days a week for 5 weeks during weeks 8-13. Patients then undergo HDR brachytherapy or IMRT once weekly during weeks 14-16.
  paclitaxel: Given IV
  carboplatin: Given IV
  external beam radiation therapy: Undergo external beam radiation therapy
  brachytherapy: Undergo HDR brachytherapy
  intensity-modulated radiation therapy: Undergo IMRT
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival
Description: One-year recurrence-free survival probability will be estimated, with 95% confidence limits based on exact methods for the binomial distribution.
Time Frame: Date of entry to date of reappearance of disease, assessed at 1 year
Population: Recurrence-free survival data was not collected/aggregated and therefore not analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Every 3 months for the first 2 years and every 6 months for the next 3 years. Up to 5 years total as described in Section 7.4 of the Study Protocol.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiotherapy)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Radiotherapy) (N=11)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) — Both Grade 1 events
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) — Grade 1
Urinary Tract Infection (Infections and infestations) | 1 (1) — Grade 2
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Grade 1
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Verbatim term Neutropenia. Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) — Grade 1
Papulopustular Rash (Infections and infestations) | 1 (1) — Grade 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Leukopenia (Blood and lymphatic system disorders) | 1 (2) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT01367301/Prot_SAP_000.pdf